CLINICAL TRIAL: NCT00640640
Title: The Effect of Intravitreal Bevacizumab & Ranibizumab on Ocular Pulse Amplitude in Neovascular Age Related Macular Degeneration
Brief Title: The Effects of Bevacizumab and Ranibizumab on Ocular Pulse Amplitude in Neovascular Age Related Macular Degeneration (AMD)
Acronym: AMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Ehud Rechtman MD, Goldschleger Eye Institute, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SHEBA-07-4739-ER-CTIL
Record Dates: First submitted 2008-02-24; First posted 2008-03-21 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2008-03

CONDITIONS: Neovascular Age Related Macular Degeneration
Keywords: IOP; OPA; AMD; bevacizumab; ranibizumab; choroidal blood flow; DCT; Ocular Pulse Amplitude change following anti VEGF; Ocular Pulse Amplitude
MeSH Terms: interventions — Ranibizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): All study patients will be evaluated in a similar way
  Interventions: Device: Pascal Dynamic Contour Tonometer; Drug: Ranibizumab; Drug: Bevacizumab

INTERVENTIONS:
Device: Pascal Dynamic Contour Tonometer — Pascal Dynamic Contour Tonometer is an ocular device that is able to safely measure the intraocular pressure and the ocular pulse amplitude
  Other Names: Pascal Dynamic Contour Tonometer = Pascal DCT
Drug: Ranibizumab — measure the effect of intravitreal 0.5mg/0.05ml ranibizumab on the intraocular pressure and ocular pulse amplitude with the Pascal Dynamic Contour Tonometer
  Other Names: Lucentis
Drug: Bevacizumab — measure the effect of intravitreal 1.25mg/0.05ml bevacizumab on the intraocular pressure and ocular pulse amplitude with the Pascal Dynamic Contour Tonometer
  Other Names: Avastin

SUMMARY:
One concern about repeated intravitreal injections of bevacizumab (Avastin) and ranibizumab (Lucentis) in wet age related macular degeneration, is that in addition to blocking the proteins that triggers the development and proliferation of abnormal vessels in the center of the retina, they may also result in changes in the normal vessels that feeds the outer part of the retina.

Small vessels with fenestrations (such as those that feed the outer part of the retina, which are called choriocapillaris) appear to be especially sensitive to this protein (called vascular endothelial growth factor, VEGF) withdrawal.

It is estimated that global blood flow in the vascular layer under the retina (called choroid) may be indirectly assessed by measuring the amplitude of the ocular pulsation (the pressure inside the eye change according to the cardiac cycle, similar to the change in blood pressure) which is called Ocular Pulse Amplitude (OPA). The Pascal Dynamic Contour Tonometer (Pascal DCT) is a new tonometer (a device which measures the pressure within the eye) designed to measure intraocular pressure and ocular pulse amplitude.

No published study has yet assessed the effect of bevacizumab (Avastin) or ranibizumab (Lucentis) treatment for wet AMD (or on any other retinal disease) on OPA. This is our aim in this pilot study, in which we will measure the pressure within the eye just prior to bevacizumab/Ranibizumab treatment, followed by repeated measurements a week and a month after the treatment.

For this purpose, up to 60 patients with wet AMD will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female in the ages of 50 year or older
2. Willing and able to sign an inform consent

Exclusion Criteria:

1. Any history, signs or symptoms of any retinal or optic nerve disease, except AMD and mild hypertensive retinopathy
2. In the presently bevacizumab/ranibizumab treated eye, prior PDT and/or intravitreal Kenalog, during the last 3 months.
3. History of ocular surgery with the following exception: extra capsular cataract extraction with implantation of a posterior chamber intra-ocular lens.
4. History of ocular laser treatment, with the following exceptions: Posterior capsulotomy following cataract surgery.
5. Cataract or other media opacity precluding adequate fundus visualization of both eyes

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-12 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Ocular pulse pressure (OPA)a week and month after intravitreal bevacizumab/ranibizumab, as compare to baseline OPA, just prior to treatment | One month for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Rechtman, MD, Principal Investigator — Sheba Medical Center
Locations (2):
- University Hospitals Leuven, Leuven, Belgium
- Goldschleger Eye Institute Sheba Medical Center, Ramat Gan, Israel